CLINICAL TRIAL: NCT00169416
Title: Clinical Evaluation of Valaciclovir Hydrochloride: 256U87 in Patients With Chickenpox - Open Uncontrolled Study.
Brief Title: Evaluation Of Valaciclovir In Patients With Chickenpox
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS2101951
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Varicella
Keywords: chicken pox; varicella; VZV; pharmacokinetics
MeSH Terms: conditions — Chickenpox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: valaciclovir HCl granules

SUMMARY:
This study will assess the safety and efficacy, and the pharmacokinetics of aciclovir and valaciclovir in children with chickenpox following oral administration of valaciclovir, for the purpose of seeking approval of valaciclovir HCl for the treatment of chickenpox.

ELIGIBILITY:
Inclusion criteria:

* Subjects aged 1 year to less than 12 years with a clinical diagnosis of chickenpox within 48 hours of the onset of the rash.

Exclusion criteria:

* History of hypersensitivity reactions.
* Impaired hepatic or renal function.
* Gastrointestinal dysfunction.
* Serious underlying disease.
* Weigh over 40kg.
* Vaccinated for chickenpox.

Ages: 1 Year to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2005-03; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Plasma aciclovir concentrations approximately 1 - 2 hours post-dose, and/or 1, 2, 4 and 6 hours following administration of the valaciclovir HCl granules 25mg/kg -dose.

SECONDARY OUTCOMES:
Plasma valaciclovir concentrations approximately 1 - 2 hours post-dose, and/or 1, 2, 4 and 6 hours following administration of the valaciclovir HCl granules 25mg/kg -dose.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline